CLINICAL TRIAL: NCT04200664
Title: Clinical and Imaging Biomarkers of Audiovestibular Function in Infratentorial Superficial Siderosis
Brief Title: Audiovestibular Function in Infratentorial Superficial Siderosis
Acronym: AViSS
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Collaborators: NIHR UCLH Biomedical Research Centre (BRC) (Unknown); Bernice Bibby Research Trust (Unknown)
Responsible Party: Sponsor
Other Study IDs: 121603
Record Dates: First submitted 2019-12-10; First posted 2019-12-16 (Actual); Results first posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Siderosis; Neurological Disorder; Rare Diseases; Age Related Hearing Loss; Presbycusis
Keywords: Superficial siderosis, infratentorial; Nervous system diseases; Hearing loss; Hearing tests; Auditory pathways; Vestibulocochlear nerve; Ataxia; Vestibular function tests; Biomarkers; Central nervous system
MeSH Terms: conditions — Siderosis; Nervous System Diseases; Rare Diseases; Presbycusis; Hearing Loss; Ataxia | interventions — Smell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva sampling to biobank the DNA for genetic analysis (siderosis group participants only). The samples will be labelled with a unique study code and will not contain identifiable information.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Siderosis (iSS) group: participants with a known diagnosis of infratentorial superficial siderosis (defined using standardised radiological criteria) confirmed by a consultant neurologist with expertise in this condition at University College London Hospitals National Health Service (NHS) Foundation Trust
  Interventions: Diagnostic Test: Hearing assessment; Diagnostic Test: Vestibular/balance assessment; Other: Quality of life assessment; Diagnostic Test: Olfactory (smell) function testing; Genetic: DNA bio-banking
- Age-related hearing loss (ARHL) group: participants with age-related hearing loss (as identified from participant's clinical history and examination, with hearing thresholds confirmed on a pure-tone audiogram)
  Interventions: Diagnostic Test: Hearing assessment; Other: Quality of life assessment
- Control group: participants with no known or previously reported hearing loss (as identified from participant's clinical history and examination, with hearing thresholds confirmed on a pure-tone audiogram)
  Interventions: Diagnostic Test: Hearing assessment; Other: Quality of life assessment

INTERVENTIONS:
Diagnostic Test: Hearing assessment — All study participants will undergo hearing tests, including hearing-specific questionnaires
Diagnostic Test: Vestibular/balance assessment — Siderosis group participants will undergo vestibular/balance tests, including gait assessment and balance-specific questionnaires
  Groups: Siderosis (iSS) group
Other: Quality of life assessment — All study participants will be asked to complete a set of quality of life questionnaires
Diagnostic Test: Olfactory (smell) function testing — Siderosis group participants will undergo a formal smell identification testing by means of self-administered smell chart to identify the revealed scents
  Groups: Siderosis (iSS) group
Genetic: DNA bio-banking — Siderosis group participants will be asked to provide a saliva sample for DNA bio-banking
  Groups: Siderosis (iSS) group

SUMMARY:
One in six people in the United Kingdom and over 400 million people worldwide have disabling hearing loss. This figure will double by 2050 as predicted by the World Health Organisation. There is an urgent need to improve our knowledge regarding hearing loss, its underlying mechanisms, optimal diagnostic modalities, reliable and accurate functional and imaging biomarkers.

A less-well studied condition associated with progressive hearing loss is infratentorial superficial siderosis (iSS). It results from iron deposition along the surfaces of brain structures which control hearing and balance. It is currently considered uncommon, but may well be under-recognised and therefore under-reported. Despite its severity, our current understanding of its impact on the hearing (auditory) and balance (vestibular) functions is limited, and this has an adverse impact on the treatment offered to these patients. Additionally, iSS patients have been reported to have cognitive impairment yet literature reports of cognitive assessment in iSS are few. The cognitive dysfunction may be specific to iSS or due to progressive hearing impairment or a combination of both, and further studies are required to establish this. Olfaction is also known to be affected in patients with iSS yet is rarely reported in the literature.

Due to the significant morbidity and progressive nature, there is a clear need to improve our understanding of the audiovestibular dysfunction resulting from iSS.

The aim of this study is to comprehensively assess audiovestibular function in iSS compared to age-related hearing loss and the controls/normative data and as a means to quantify deficits for monitoring disease progression and response to treatment, to assess the impact on the quality of life, to analyse clinically-obtained data (including imaging, cognitive and laboratory data), and correlate these with functional findings in iSS.

DETAILED DESCRIPTION:
This study focuses on a rare condition called infratentorial superficial siderosis (iSS)-a disease where iron gradually accumulates in the superficial layers of the brain and spinal cord. Over time, this buildup can damage the nerves responsible for hearing and balance amongst others, leading to symptoms like progressive hearing loss, dizziness, and problems with coordination. iSS has not been well studied in the past. The hearing and balance function in persons with iSS has been described as variable - meaning, there has not been a specific pattern of hearing loss or imbalance or dizziness that can be associated with iSS. The studies to date have been with small groups of patients but mainly case reports.

The aim of the AVISS study has been to address this gap in the knowledge. This study investigates how iSS affects hearing, balance, and even sense of smell by studying three groups of people:

1. People with iSS, who already have hearing and balance problems.
2. People with age-related hearing loss, to compare how hearing declines over time.
3. People with normal hearing, serving as a control group.

The study will take place over three years, using a range of tests to assess hearing and balance:

* Hearing tests like pure tone audiometry, speech-in-noise assessments, and auditory brainstem response.
* Balance tests such as vestibular evaluations, gait assessments, and head impulse testing.
* Olfactory (smell) tests, since iSS might also affect sensory perception. By collecting this data, the study aims to improve how iSS is diagnosed, identify better rehabilitation methods, and explore new treatment options for those affected.

The study is funded by NIHR UCLH Biomedical Research Centre and the Bernice Bibby Research Trust, ensuring experts have the resources needed to make meaningful discoveries. Ultimately, the goal is to help doctors recognize iSS earlier, support affected individuals more effectively and improve their overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Siderosis group: adults (male and female) of 18+ years old with a known diagnosis of iSS (defined using standardised radiological criteria) confirmed by a consultant neurologist with expertise in this condition at University College London Hospitals National Health Service (NHS) Foundation Trust
* Age-related hearing loss (ARHL) group: adults (male and female) of 18+ years old with ARHL
* Control group: adults (male and female) of 18+ years old with no previous diagnosis of hearing loss or no known neurological disorder (including iSS) that affects hearing, with the aim to recruit such participants of 50 years of age and above; however, should difficulty with the recruitment of such participants arise, participants of 18 years of age and above will be invited to participate in the study.

Exclusion Criteria:

* All groups: individuals younger than 18 years old; individuals with a physical or mental impairment that prevents the potential participant from giving informed consent or undergoing the hearing and/or vestibular assessment;
* Siderosis group: individuals with no prior diagnosis of iSS
* Age-related hearing loss (ARHL) group: individuals with no previous diagnosis of ARHL or with a diagnosis of hearing loss of aetiology other than age-related; individuals with a history of exposure to high-intensity noise or ototoxic drugs or evidence of middle ear disease/dysfunction or family history of non age-related hearing loss;
* Control group: individuals with a known history of hearing loss (of any cause) or with a known neurological disorder that affects their hearing; individuals with history of exposure to high-intensity noise or ototoxic drugs or evidence of middle ear disease or family history of non age-related hearing loss;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Three groups of participants will be recruited into the study (as defined by the eligibility criteria): a) participants with a known diagnosis of iSS (siderosis group); b) participants with age-related hearing loss (ARHL group); c) participants with no previous history of hearing loss (control group).
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2021-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doris-Eva Bamiou, Professor, Principal Investigator — UCL Ear Institute; UCLH NHS Foundation Trust, UK; David J Werring, Professor, Principal Investigator — Stroke Research Centre UCL IoN; UCLH NHS Foundation Trust, UK
Locations (2):
- United Kingdom (2):
  - UCL Ear Institute, London
  - University College London Hospitals NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No
The anonymised participant-level dataset and statistical code for generating the results will not be publicly available.

REFERENCES:
- [Background] Wilson D, Chatterjee F, Farmer SF, Rudge P, McCarron MO, Cowley P, Werring DJ. Infratentorial superficial siderosis: Classification, diagnostic criteria, and rational investigation pathway. Ann Neurol. 2017 Mar;81(3):333-343. doi: 10.1002/ana.24850. Epub 2017 Jan 28. PMID 28019651
- [Background] Fearnley JM, Stevens JM, Rudge P. Superficial siderosis of the central nervous system. Brain. 1995 Aug;118 ( Pt 4):1051-66. doi: 10.1093/brain/118.4.1051. PMID 7655881
- [Background] Koeppen AH, Dickson AC, Chu RC, Thach RE. The pathogenesis of superficial siderosis of the central nervous system. Ann Neurol. 1993 Nov;34(5):646-53. doi: 10.1002/ana.410340505. PMID 8239558
- [Background] Kumar N. Superficial siderosis: associations and therapeutic implications. Arch Neurol. 2007 Apr;64(4):491-6. doi: 10.1001/archneur.64.4.491. PMID 17420310
- [Background] IWANOWSKI L, OLSZEWSKI J. The effects of subarachnoid injections of iron-containing substances on the central nervous system. J Neuropathol Exp Neurol. 1960 Jul;19:433-48. doi: 10.1097/00005072-196007000-00010. No abstract available. PMID 14406175
- [Background] Posti JP, Juvela S, Parkkola R, Roine S. Three cases of superficial siderosis of the central nervous system and review of the literature. Acta Neurochir (Wien). 2011 Oct;153(10):2067-73. doi: 10.1007/s00701-011-1116-0. Epub 2011 Aug 7. PMID 21822983
- [Background] Sydlowski SA, Cevette MJ, Shallop J. Superficial siderosis of the central nervous system: phenotype and implications for audiology and otology. Otol Neurotol. 2011 Aug;32(6):900-8. doi: 10.1097/MAO.0b013e31822558a9. PMID 21730883
- [Background] Offenbacher H, Fazekas F, Schmidt R, Kapeller P, Fazekas G. Superficial siderosis of the central nervous system: MRI findings and clinical significance. Neuroradiology. 1996 May;38 Suppl 1:S51-6. doi: 10.1007/BF02278119. PMID 8811680
- [Background] Sydlowski SA, Levy M, Hanks WD, Clark MD, Ackley RS. Auditory profile in superficial siderosis of the central nervous system: a prospective study. Otol Neurotol. 2013 Jun;34(4):611-9. doi: 10.1097/MAO.0b013e3182908c5a. PMID 23670174
- [Background] Vibert D, Hausler R, Lovblad KO, Schroth G. Hearing loss and vertigo in superficial siderosis of the central nervous system. Am J Otolaryngol. 2004 Mar-Apr;25(2):142-9. doi: 10.1016/j.amjoto.2003.10.001. PMID 14976664
- [Background] Takeda T, Kawashima Y, Hirai C, Makabe A, Ito T, Fujikawa T, Yamamoto K, Maruyama A, Tsutsumi T. Vestibular Dysfunction in Patients With Superficial Siderosis of the Central Nervous System. Otol Neurotol. 2018 Jul;39(6):e468-e474. doi: 10.1097/MAO.0000000000001844. PMID 29889788
- [Background] Pribitkin EA, Rondinella L, Rosenberg Si, Yousem DM. Superficial siderosis of the central nervous system: an underdiagnosed cause of sensorineural hearing loss and ataxia. Am J Otol. 1994 May;15(3):415-8. PMID 8579152
- [Background] Kwartler JA, De La Cruz A, Lo WW. Superficial siderosis of the central nervous system. Ann Otol Rhinol Laryngol. 1991 Mar;100(3):249-50. doi: 10.1177/000348949110000315. No abstract available. PMID 2006825
- [Background] van Harskamp NJ, Rudge P, Cipolotti L. Cognitive and social impairments in patients with superficial siderosis. Brain. 2005 May;128(Pt 5):1082-92. doi: 10.1093/brain/awh487. Epub 2005 Mar 23. PMID 15788543
- See also: WHO global estimates on prevalence of hearing loss — https://www.who.int/health-topics/hearing-loss#tab=tab_2

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 90 anticipated participants, only 11 participants were recruited to the study - into the Siderosis group. Participants were not recruited into the non siderosis groups (ie Age-Related Hearing Loss group and Control group) due COVID19 restrictions at the time of the study, which impacted significantly on recruitment opportunities and dramatically reduced the participant number in the study.
Pre-assignment Details: There were limited opportunities to recruit participants into study, (we anticipated 30 participants in each group). The apparent discrepancy between the anticipated recruitment number and the actual number of participants across all groups was due to COVID-19 pandemic and social restrictions placed. Subsequent easing off of the restrictions allowed to recruit 11 participants (from November 2019 to July 2021) but study-related time constraints did not allow to proceed with further recruitment.
Groups:
- Age-related Hearing Loss (ARHL) Group: Age-Related Hearing Loss group not recruited due to the impact of COVID19 on recruitment opportunities.
- Control Group: Control group not recruited due to the impact of COVID19 on recruitment opportunities.
Period: Overall Study
Arm/Group | Siderosis (iSS) Group | Age-related Hearing Loss (ARHL) Group | Control Group
Started | 11 | 0 | 0
Completed | 10 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Individuals with known/confirmed diagnosis of infratentorial classical superficial siderosis under the care of clinical team at the UCLH NHS Foundation Trust, UK.
Arm/Group | Siderosis (iSS) Group
Number analyzed (Participants) | 10
Age, Customized [Mean (Standard Deviation); unit: years] | 52.5 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Hearing Evaluation - Pure Tone Audiometry
Description: Clinical audiological (hearing) tests were performed to assess hearing function. The hearing tests included psychophysical, physiological and electrophysiological measures, (pure-tone audiometry, tympanometry, auditory brainstem responses and acoustic reflexes). The tests were perfomed in line with the procedure guidelines by the British Society of Audiology (www.thebsa.org.uk). The mean value of pure-tone audiometric thresholds for both ears measured in decibel hearing level (as described in the guidelines by the British Society of Audiology) was calculated and reported. Other parameters were reported as normal or abnormal (in at least one ear) or inconclusive.
Time Frame: Baseline visit
Population: Participants with known diagnosis of infratentorial superficial siderosis.
Measure: Mean (Standard Deviation); unit: decibel hearing level
Arm/Group | Siderosis (iSS) Group
Number analyzed (Participants) | 11
decibel hearing level | 57.3 (39.9)

2. Primary Outcome: Vestibular/Balance Evaluation
Description: Clinical vestibular and balance tests were performed to assess vestibular/balance function.
Time Frame: Baseline visit
Population: Vestibular tests included video head impulse test, oculomotor and rotatory chair testing using video or electronystagmography; bithermal calorics, ocular and cervical vestibular evoked myogenic potentials. The results are presented as normal if bilateral or unilateral normal findings;
Measure: Count of Participants; unit: Participants
Arm/Group | Siderosis (iSS) Group
Number analyzed (Participants) | 10
Participants
  Video head impulse test: Abnormal | 6
  Video head impulse test: Normal | 1
  Video head impulse test: Not tested | 3
  Video- electro-nystagmography (oculomotor; rotatory chair) - central vestibular assessment: Abnormal | 9
  Video- electro-nystagmography (oculomotor; rotatory chair) - central vestibular assessment: Normal | 1
  Video- electro-nystagmography (oculomotor; rotatory chair) - central vestibular assessment: Not tested | 0
  Video- electronystagmography (oculomotor; rotatory chair) - peripheral vestibular assessment: Abnormal | 7
  Video- electronystagmography (oculomotor; rotatory chair) - peripheral vestibular assessment: Normal | 3
  Video- electronystagmography (oculomotor; rotatory chair) - peripheral vestibular assessment: Not tested | 0
  Bithermal calorics: Abnormal | 1
  Bithermal calorics: Normal | 2
  Bithermal calorics: Not tested | 7
  ocular Vestibular Evoked Myogenic Potentials: Abnormal | 0
  ocular Vestibular Evoked Myogenic Potentials: Normal | 9
  ocular Vestibular Evoked Myogenic Potentials: Not tested | 1
  cervical Vestibular Evoked Myogenic Potentials: Abnormal | 3
  cervical Vestibular Evoked Myogenic Potentials: Normal | 7
  cervical Vestibular Evoked Myogenic Potentials: Not tested | 0

3. Primary Outcome: Hearing Evaluation - Auditory Brainstem Responses/Acoustic Reflexes
Description: as for outcome 1
Time Frame: Baseline visit
Population: Results for psychophysical, physiological/electrophysiological measures (units: participants); normal if bilateral or unilateral normal findings; Auditory brainstem responses were recorded as normal, abnormal or inconclusive
Measure: Count of Participants; unit: Participants
Arm/Group | Siderosis (iSS) Group
Number analyzed (Participants) | 11
Participants
  Abnormal | 5
  Inconclusive | 2
  Not performed | 4

4. Primary Outcome: Hearing Evaluation - Tympanogram
Description: as for outcome 1
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Siderosis (iSS) Group
Number analyzed (Participants) | 11
Participants
  Abnormal | 0
  Normal | 11

5. Primary Outcome: Hearing Evaluation - Otoacoustic Emissions
Description: as for outcome 1
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Siderosis (iSS) Group
Number analyzed (Participants) | 11
Participants
  Present | 3
  Absent | 3
  Not performed | 5

6. Primary Outcome: Hearing Evaluation - Listening in Spatialised Sentences Noise Test
Description: Clinical audiological (hearing) tests were performed to assess hearing function. The hearing tests included psychophysical, physiological and electrophysiological measures, (pure-tone audiometry, tympanometry, auditory brainstem responses and acoustic reflexes). The tests were perfomed in line with the procedure guidelines by the British Society of Audiology (www.thebsa.org.uk). The mean value of pure-tone audiometric thresholds for both ears measured in decibel hearing level (as described in the guidelines by the British Society of Audiology) was calculated and reported. Other parameters were reported as normal or abnormal (in at least one ear) or inconclusive. Cameron S, Dillon H. The listening in spatialized noise-sentences test (LISN-S): comparison to the prototype LISN and results from children with either a suspected (central) auditory processing disorder or a confirmed language disorder. J Am Acad Audiol. 2008 May;19(5):377-91.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Siderosis (iSS) Group
Number analyzed (Participants) | 11
Participants
  Abnormal | 4
  Normal | 1
  Not tested | 6

7. Secondary Outcome: Correlation Between Clinically Obtained Imaging (Siderosis Group Participants) and the Hearing and Balance Assessment Results
Description: Siderosis group participants underwent formal imaging procedures as part of their clinical care pathway. The imaging results were reviewed with the results obtained from hearing and vestibular/balance assessments. All participants had MRI Brain, as part of their clinical care pathway; susceptibility-weighted images were reviewed to identify the appearance of superficial siderosis, in keeping with the radiological diagnostic criteria (Reference: Wilson et al, 2017).
Time Frame: Baseline visit
Measure: Count of Participants; unit: Participants
Arm/Group | Siderosis (iSS) Group
Number analyzed (Participants) | 10
Participants
  Superior cerebellar vermis: Hypointense signal consistent with superficial siderosis observed | 10
  Superior cerebellar vermis: Hypointense signal consistent with superficial siderosis not observed | 0
  Cerebellar folia: Hypointense signal consistent with superficial siderosis observed | 10
  Cerebellar folia: Hypointense signal consistent with superficial siderosis not observed | 0
  Midbrain: Hypointense signal consistent with superficial siderosis observed | 10
  Midbrain: Hypointense signal consistent with superficial siderosis not observed | 0
  Pons: Hypointense signal consistent with superficial siderosis observed | 9
  Pons: Hypointense signal consistent with superficial siderosis not observed | 1
  Medulla: Hypointense signal consistent with superficial siderosis observed | 9
  Medulla: Hypointense signal consistent with superficial siderosis not observed | 1
  8th cranial nerve (unilateral or bilateral): Hypointense signal consistent with superficial siderosis observed | 9
  8th cranial nerve (unilateral or bilateral): Hypointense signal consistent with superficial siderosis not observed | 1
  Supratentorial extension: Hypointense signal consistent with superficial siderosis observed | 10
  Supratentorial extension: Hypointense signal consistent with superficial siderosis not observed | 0
  Sylvian fissures: Hypointense signal consistent with superficial siderosis observed | 9
  Sylvian fissures: Hypointense signal consistent with superficial siderosis not observed | 1

8. Secondary Outcome: Correlation Between Clinically Obtained Results of Cognitive Function Assessment (Siderosis Group Participants) and the Hearing and Balance Assessments
Description: Siderosis group participants underwent a formal neuro-cognitive assessment as part of their clinical care pathway. The results of this clinical assessment were reviewed to determine if an association exists between the cognitive assessment results and the results obtained from hearing and vestibular/balance assessments performed during the study. A formal neuro-cognitive assessment was performed using the Wechsler Adult Intelligence Scale test. Cognitive impairment in a domain was defined as scoring at or below the fifth percentile on any one test in that domain.
Time Frame: Baseline visit
Measure: Count of Participants; unit: Participants
Arm/Group | Siderosis (iSS) Group
Number analyzed (Participants) | 7
Participants
  Participants who underwent neurocognitive assessment | 7
  Executive function abnormal | 5
  Visual memory abnormal | 5
Statistical Analysis 1: Comparison: Siderosis (iSS) Group; Test type: Other — Kendall tau b correlation analysis test was performed between the number of cognitive domains affected and the both ears 3-frequency pure tone average (at 0.5/1/2kHz) or both ears 4-frequency pure tone average (at 0.5/1/2/4kHz); p = 0.176, Kendall tau-b; Kendall tau b non-parametric correlation analysis was performed; Kendall Tau-b = 0.462

9. Secondary Outcome: Smell Identification Test
Description: University of Pennsylvania Smell Identification Test (UPSIT, British version) was performed (siderosis group participants) to assess their olfactory function. UPSIT is a forced-choice 40-item self-administered test. The scores are calculated using manufacturer's answer key as the sum of correct answers (maximum best = 40, minimum score 6; anosmia <19(males, females); normosmia >33 (males) and >34 (females)), and compared to the age- and gender-matched norms. The scores are also grouped into categories (ranging from normosmia to anosmia), with higher scores indicating better olfactory function.
Time Frame: Baseline visit
Measure: Mean (Standard Deviation); unit: UPSIT score
Arm/Group | Siderosis (iSS) Group
Number analyzed (Participants) | 10
UPSIT score | 25.5 (7.8)

ADVERSE EVENTS:
Time Frame: Up to one hour at baseline
Description: This was an observational study to assess auditory, vestibular, and olfactory functions in individuals with a known diagnosis of infratentorial superficial siderosis. No adverse events or serious adverse events were recorded during the study.
Arm/Group | Siderosis (iSS) Group
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

LIMITATIONS AND CAVEATS:
The tests were performed at baseline only. The major limitation to the study was the impact of COVID-19 pandemic on participant recruitment, availability of testing facilities and overall social restricions that were in place during the COVID-19 pandemic while the study was open.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/64/NCT04200664/Prot_SAP_000.pdf